CLINICAL TRIAL: NCT07297199
Title: A Phase 1, Randomized, Open-Label, Single-Dose, Crossover, Bioequivalence Study of Omaveloxolone Tablets for Oral Suspension Versus Capsules in Healthy Adult Participants
Brief Title: A Study to Learn How the Body Processes BIIB141 (Omaveloxolone) When Taken as a Capsule or as a Tablet Dissolved in Liquid, and to Learn About Its Safety in Healthy Adults Ages 18 to 55
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 296HV102
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — omaveloxolone

STUDY DESIGN:
Intervention Model Description: This 2-way crossover study will be conducted in 2 periods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence AB (Experimental): Participants will receive treatment A (omaveloxolone capsule orally) on Day 1 followed by treatment B (omaveloxolone TOS) on Day 15.
  Interventions: Drug: Omaveloxolone
- Treatment Sequence BA (Experimental): Participants will receive treatment B (omaveloxolone TOS) on Day 1 followed by treatment A (omaveloxolone capsule orally) on Day 15.
  Interventions: Drug: Omaveloxolone

INTERVENTIONS:
Drug: Omaveloxolone — Administered orally
  Other Names: BIIB141; SKYCLARYS

SUMMARY:
In this study, researchers will learn more about BIIB141, also known as omaveloxolone or SKYCLARYS®. This drug has been approved, or made available for doctors to prescribe, for people with Friedrich's Ataxia (FA) who are at least 16 years old. Currently, BIIB141 is taken by mouth as capsules or capsule contents sprinkled over applesauce. But, there may be some people who have trouble swallowing capsules. In this study, the main goal was to learn if BIIB141 is processed similarly in the body of healthy adults when taken as tablets that dissolve in liquid compared to the currently available capsules.

The main question researchers want to answer in this study is :

• How does the body process BIIB141 when taken as a tablet dissolved in liquid compared to capsules?

Researchers will also learn more about:

* How many participants have adverse events during the study. An adverse event is a health problem that may or may not be caused by the study drug.
* If there are any changes in the participants' overall health during the study.

This study will be done as follows:

* Participants will be screened to check if they can join the study. The screening period will be up to 28 days, after which participants will check into their study research center.
* Participants will stay at the study research center for about 30 days.
* This is an "open label" study. In this kind of study, the participants, study doctor, and site staff know which study drug the participant is taking. In this study, all participants will take BIIB141.
* This study also has a "crossover" design. This means that all of the participants will take BIIB141, once as a tablet that dissolves in liquid and once as a capsule. But the order in which the participants take them will be different. There will be a break of about 14 days between the 2 doses.
* Throughout the study, researchers will take participants' blood and urine samples. Researchers will also do other tests to check the participants' overall health and will ask participants how they are feeling.
* Each participant will be in the study for up to 57 days.

DETAILED DESCRIPTION:
The primary objective of the study is to assess the bioequivalence (BE) of omaveloxolone tablets for oral suspension (TOS) compared to capsules in healthy adult participants. The secondary objective of the study is to assess the safety and tolerability of a single dose of omaveloxolone when administered as TOS or capsule in healthy adult participants.

ELIGIBILITY:
Key Inclusion Criteria:

* All female participants of childbearing potential must have negative results for pregnancy tests as follows:

  1. At screening, based on a serum sample obtained within 28 days prior to initial study drug administration; and
  2. Prior to dosing, based on a serum sample obtained on Study Day -1.
* Body Mass Index (BMI) at screening between 18 and 32 kilograms per meter square (kg/m^2), inclusive.
* Participants must be in good health.

Key Exclusion Criteria:

* History of any clinically significant cardiac, endocrine, gastrointestinal, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, or renal disease, or other major disease, as determined by the Investigator.
* Clinically significant, as determined by the Investigator, 12-lead electrocardiogram (ECG) abnormalities.
* History of, or positive test result for human immunodeficiency virus (HIV).
* History of hepatitis C infection or positive test result at Screening for hepatitis C virus antibody (HCV Ab).
* Current hepatitis B infection [defined as positive for hepatitis B surface antigen (HBsAg) and/or total hepatitis B core antibody (anti-HBc)]. Participants with immunity to hepatitis B from previous natural infection (defined as negative HBsAg, positive anti-HBc, and positive anti-HBs) or vaccination (defined as negative HBsAg, negative anti-HBc, and positive anti-HBs) are eligible to participate in the study.
* Chronic, recurrent, or serious infection (e.g., pneumonia, septicemia), as determined by the Investigator, within 90 days prior to Screening or between Screening and Day -1.
* Prior exposure to the study treatment.
* Any clinically significant abnormal laboratory test value as determined by the Investigator, as Screening or Day-1.

NOTE: Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2026-04-17 (Estimated); Study Completion 2026-04-17 (Estimated)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Omaveloxolone | Pre-dose and at multiple timepoints post-dose up to Day 29
Area Under the Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Omaveloxolone | Pre-dose and at multiple timepoints post-dose up to Day 29

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to end of study (up to Day 29)
Number of Participants With Clinically Significant Change From Baseline in Laboratory Abnormalities | From Day 1 up to end of study (up to Day 29)
Number of Participants With Change From Baseline in Clinically Relevant Vital Sign Abnormalities | From Day 1 up to end of study (up to Day 29)
Number of Participants With Change From Baseline in Clinically Relevant Electrocardiogram (ECG) Abnormalities | From Day 1 up to end of study (up to Day 29)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Trialmed formerly PPD, Austin Clinical Research Unit, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/